CLINICAL TRIAL: NCT00112515
Title: Pilot Study Evaluating the Safety and Efficacy of Modafinil in Improving Fatigue, Mood, Cognitive Ability, Functional Status, and Quality of Life of Cancer Patients
Brief Title: Modafinil in Treating Fatigue in Patients With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000432953; UVACC-HIC-10951; UVACC-30603
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2006-05

CONDITIONS: Cognitive/Functional Effects; Depression; Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: depression; cognitive/functional effects; fatigue; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Depression; Fatigue | interventions — Modafinil; Mental Status and Dementia Tests; Psychiatric Rehabilitation

INTERVENTIONS:
Drug: modafinil
Procedure: cognitive assessment
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Modafinil may help relieve fatigue and improve quality of life in patients with cancer.

PURPOSE: This clinical trial is studying how well modafinil works in treating fatigue in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of modafinil in cancer patients.
* Determine the efficacy of this drug, in terms of improving fatigue, in these patients.

Secondary

* Determine the efficacy of this drug, in terms of improving mood, cognitive ability, functional status, and quality of life, in these patients.

OUTLINE: This is a nonrandomized, pilot study.

Patients receive oral modafinil once daily for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients may receive additional modafinil at the discretion of the physician.

Fatigue, mood, cognition, functional status, and quality of life are assessed at baseline and in weeks 2 and 4.

After completion of study treatment, patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 26 patients will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Brief Fatigue Inventory score ≥ 4

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 1-3

Life expectancy

* At least 2 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No history of left ventricular hypertrophy
* No history of ischemic ECG changes
* No history of chest pain
* No history of arrhythmia
* No history of other clinically significant manifestations of mitral valve prolapse in association with CNS stimulant use

Other

* Not pregnant or nursing
* Negative pregnancy test
* Thyroid stimulating hormone normal
* No known hypersensitivity to modafinil
* No history of psychotic disorder and/or active psychosis
* No history of any chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation or compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent thalidomide allowed

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Concurrent narcotics, phenothiazines, or benzodiazepines allowed
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02

PRIMARY OUTCOMES:
Safety, in terms of adverse events and dose-limiting toxicity, as measured by NCI CTC v2.0 at up to 4 weeks after the start of treatment
Fatigue as measured by Brief Fatigue Inventory at 2 and 4 weeks after the start of treatment

SECONDARY OUTCOMES:
Mood as measured by Hamilton Rating Scale for Depression at 2 and 4 weeks after the start of treatment
Cognitive ability (i.e., memory, fine motor control, fluency, general mental ability, & delayed memory) by Hopkins Verbal Learning Test at 2 and 4 weeks after start of treatment
Cognitive ability (i.e., memory, fine motor control, fluency, general mental ability, & delayed memory) by Grooved Pegboard Test at 2 and 4 weeks after start of treatment
Cognitive ability (i.e., memory, fine motor control, fluency, general mental ability, & delayed memory) by Controlled Oral Word Association Test from the Multilingual Aphasia Examination at 2 and 4 weeks after start of treatment
Cognitive ability (i.e., memory, fine motor control, fluency, general mental ability, & delayed memory) by Trail Making Test A and B at 2 and 4 weeks after start of treatment
Cognitive ability (i.e., memory, fine motor control, fluency, general mental ability, & delayed memory) by Recall and Recognition of Word List encoded from the Hopkins Verbal Learning Test at 2 and 4 weeks after start of treatment
Functional status as measured by Barthel Index and ECOG performance status at 2 and 4 weeks after the start of treatment
Quality of life as measured by Functional Assessment of Cancer Therapy-Br at 2 and 4 weeks after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Blackhall, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States